CLINICAL TRIAL: NCT05719610
Title: Effects of Cawthorne Cooksey Exercises on Balance and Quality of Life in Children With Hearing Deficits
Brief Title: Effects of Cawthorne Cooksey Exercises on Balance in Children With Hearing Deficits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0731
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Hearing Disorders
MeSH Terms: conditions — Hearing Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cawthorne Cooksey Exercises (Experimental)
  Interventions: Other: Cawthorne Cooksey Exercises for Balance Training
- Swiss Ball Exercises (Experimental)
  Interventions: Other: Swiss Ball Exercises

INTERVENTIONS:
Other: Cawthorne Cooksey Exercises for Balance Training — Group of Exercises used to Increase balance
  Arms: Cawthorne Cooksey Exercises
Other: Swiss Ball Exercises — Swiss Ball Exercises
  Arms: Swiss Ball Exercises

SUMMARY:
Balance and weak postural control are most common in children with severe to profound hearing deficits. Children with hearing deficits also indicate behavioral problems related to impulse control, distraction, and disability to maintain attention in the visual modality. Hearing deficit is mostly defined as a communication deficit. Although the communication deficit is an important disorder, hearing deficit co-occurs with other physical impairments such as vestibular disorders. Development and control of the posture are important prerequisites for skill motor function. Children with hearing deficits and impaired sensory organization had weak balance and motor efficiency in many fields. Various studies on motor skills in deaf children have reported deficits in balance, general dynamic coordination, visual-motor skills, ball catching ability, and some disturbances in reaction time and speed of movements. Teachers of children with hearing impairment often complain of non-coordination, clumsiness, and balance deficit in such children, preventing the child from the desired function. So the aim of the study is to determine the effects of Cawthorne Cooksey Exercises on Balance and quality of life in children with hearing deficit It will be a Randomized Controlled Trial and children fulfilling exclusion-inclusion criteria will participate in the study. They will be divided randomly into two groups, using computer generated randomization, into control group and experimental group. After performing the pre-test measurements, the control group will perform Swiss Ball Exercises for 45 minutes and the interventional group will perform Cawthorne Cooksey Training Program Swiss Ball Exercises in addition, will also perform of 45 min session three times a week for 8 weeks of training. the study subjects will be evaluated again by Pediatrics Berg Balance Scale, Four-Step Square test and Quality of life questionnaire for children to measure the quality of life. Results will be compared with the pretest measurements. Data will be analyzed by using SPSS scale windows software version 25.

DETAILED DESCRIPTION:
In children, vestibular function plays an important role in the gross motor development and postural control. Infants and children with congenitally profound hearing loss commonly suffer vestibular dysfunction in both ears, and poor balance. However, there have been very few studies have investigated the effect of exercises on balance and quality of life in children with the profound hearing deficit. The development and maintenance of balance is a multisystem process that also depends on vestibular input believe that as labyrinths and cochlea are anatomically and developmentally interrelated, there is a potentiality for vestibular impairment when the hearing mechanism is impaired.

In a study using Barany Rotary test and caloric stimulation, found that 82% of 89 children with severe acquired hearing deficits and 34% of 129 children with hereditary hearing deficits had abnormal responses to vestibular tests. Since the vestibular system activates vestibular reflex mechanisms trying to stabilize the eyes, head, and body in the space, impairment of this mechanism may affect postural sensitivity. Maturational changes in visual and proprioceptive, central nervous system processing, and coordination of motor output are responsible for the changes in postural skills observed through adolescence . From the sensory systems perspective, Infants and young children are dependent on the visual system to maintain balance; as they grow older, begin to use somatosensory and vestibular information appropriately. Between the 3 sensory inputs in children, the vestibular system seems to be the least effective in postural control.

Children with profound bilateral vestibular dysfunction present with delayed gross motor development. These children stand and walk later than their peers with typical development Difficulties in maintaining balance can lead to challenges in normal childhood activities, such as riding a bicycle or hopping. Reduced ability to participate in normal play with other children may result in social isolation. So, the mechanisms responsible for the lack of balance in children with profound hearing impairment need to be established, and holistic management including both auditory and vestibular function is needed. Sensory organization dysfunction is more prevalent in children with hearing loss and vestibular dysfunction which may result in a problem with balance. These children in situations needs an early address to their balance through balance training activities. Most children with bilateral vestibular dysfunction. These results suggest that due to multi-modal sensory interdependence, the development of visual and somatosensory effectiveness in maintaining balance is impaired secondary to vestibular dysfunction since birth. There is ample support for the efficacy of vestibular rehabilitation therapy through different exercises in adults, but very few data exist regarding its results in children.

Balance is major problem associated with vestibular system specifically in the patients with sensory neural hearing deficits. Since vestibular rehabilitation is an important factor that must be achieved for balance in hearing deficits. Cawthorne Cooksey exercises may be considered as an effective technique to gain balance and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Children with age between 7 to 12 yeas
* Children with diagnosed sensorineural hearing deficits (PTA >90db)
* Children with normal vision

Exclusion Criteria:

* Children with any orthopedic and neurological impairments
* Children taking medications that affect central nervous system
* In the case of being absent from more than two sessions, non-cooperation of the family, and the occurrence of orthopedic accidents and if diseases prevented the patient from participation

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Pediatric Berg Balance Scale | 12 weeks
  The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points

SECONDARY OUTCOMES:
Four-step square test | 12 weeks
  the FSST has been widely used in neurological populations3-5 and also in musculoskeletal conditions such as joint replacements, arthritis, osteoporosis, orthotic design for lower extremity trauma and amputees. The FSST requires a stopwatch and four single point sticks

OTHER OUTCOMES:
Quality of life questionnaire for children to measure Quality of life | 12 weeks
  This is questionnaire that is used to as a tool for the assessment for quality of life. It is a questionnaire that will be filled with the help of teacher of deaf children who is expert of sign language. It consists of questions that are easy to answer.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Khan, MS, Principal Investigator — Riphah International University
Locations (1):
- Government Secondary School of Special Education for Deaf, Main Gulberg Lahore., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No